CLINICAL TRIAL: NCT03740542
Title: A Phase III Randomized Trial of Pyloroplasty Versus No Pyloroplasty in Patients Undergoing Esophagectomy
Brief Title: Pyloroplasty Versus No Pyloroplasty in Patients Undergoing Esophagectomy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, James Luketich, Principal Investigator, University of Pittsburgh
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STUDY19020375
Record Dates: First submitted 2018-08-20; First posted 2018-11-14 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Esophagectomy
MeSH Terms: interventions — Esophagectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Esophagectomy with Pyloroplasty (Active Comparator): Esophagectomy with Pyloroplasty
  Interventions: Procedure: Esophagectomy; Procedure: Pyloroplasty
- Esophagectomy without Pyloroplasty (Experimental): Esophagectomy without Pyloroplasty
  Interventions: Procedure: Esophagectomy

INTERVENTIONS:
Procedure: Esophagectomy — Surgical removal of part of esophagus
Procedure: Pyloroplasty — pyloric drainage procedure
  Arms: Esophagectomy with Pyloroplasty

SUMMARY:
This research study is a phase III randomized trial to study the value of the addition of a pyloroplasty procedure versus no pyloroplasty procedure during the performance of esophagectomy. Pyloroplasty is a type of pyloric drainage procedure.

DETAILED DESCRIPTION:
Patients selected for enrollment in this study will be adults (18-85 years of age) that have been scheduled for exploration, and possible esophagectomy. Prior to surgery, patients will be randomized to one of two groups. Group A will have a pyloroplasty performed as part of the esophagectomy procedure. Group B will not have a pyloroplasty performed. Postoperative patient outcomes will be assessed for 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be willing to undergo esophagectomy for benign or malignant condition
* Women and men 18-85 years of age
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Stomach is used as conduit

Exclusion Criteria:

* Previous operations of the pylorus
* Previous gastric resection
* Previous gastric bypass
* Patients who are unable to tolerate surgery
* Participants may be enrolled and randomized on the study but may be excluded at the time of the surgery because of findings by the surgeon that preclude performing esophagectomy, or using stomach as a conduit or findings which preclude following the randomized arm.
* Age <18 years of age or > 85 years of age
* BMI > 50
* Liver cirrhosis or liver failure at physician's discretion

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2023-02-14 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
pneumonia | 30 days postoperatively
  Defined as meeting 3 of 5 characteristics: fever, leukocytosis, chest x-ray (CXR) with infiltrate, positive culture from sputum, or treatment with antibiotics
esophageal anastomosis leak requiring surgery | 30 days postoperatively
  Defined as a leak at the esophageal anastomosis site as evidenced by Barium Swallow Study.

SECONDARY OUTCOMES:
Mortality | 30 days
  Death within 30 days of surgery
Time to start oral diet | Up to 24 months
  Number of days from surgery to starting oral diet
Quality of life assessment by completion of SF36 Quality of Life questionnaire | Prior to esophagectomy, at the first postoperative visit, and 4, 6, and 12 months after surgery
  SF36 Quality of Life questionnaire
Gastroesophageal Reflux Disease (GERD)-Health Related Quality of Life (HRQL) measured by completion of GERD HRQL questionnaire | Prior to esophagectomy, at the first postoperative visit, and 4, 6, and 12 months after surgery.
  Gastroesophageal Reflux Disease (GERD)-Health Related Quality of Life (HRQL) questionnaire prior to esophagectomy, at the first postoperative visit, and 4, 6, and 12 months after surgery.
Dysphagia as reported by patient using the Dysphagia scale | Prior to esophagectomy, at the first postoperative visit, and 4, 6, and 12 months after surgery.
  Dysphagia scale measures swallowing difficulty on a scale of 1-5. (1=no difficulty swallowing; 2=difficulty swallowing hard solids; 3=difficulty swallowing soft solids; 4=difficulty swallowing liquids; 5=unable to swallow anything. A lower score represents a better outcome.
Nasogastric tube drainage measured in milliliters | From date of surgery until date nasogastric tube is removed or date of discharge from hospital, whichever came first, assessed up to 24 months.
  Measured in milliliters
Replacement of nasogastric tube reported as number of days from tube removal to reinsertion | Up to 24 months
  Number of days from nasogastric tube removal to reinsertion
Esophageal dilations reported as the number of esophageal dilations performed | Up to 24 months
  Number of esophageal dilations performed
Length of hospital stay | From date of surgery until the date of discharge from hospital, assessed up to 24 months.
  Number of days in hospital
Aspiration as reported on radiographic imaging | Performed when clinically indicated up to 24 months postoperatively
  Radiographic imaging reports
Gastric outlet obstruction as reported on barium swallow reports | Performed when clinically indicated up to 24 months postoperatively
  Barium swallow reports
Re-admission to hospital | Up to 24 months postoperatively
  Number of days from hospital discharge to re-admission
Unexpected return to the Operating Room | Up to 24 months postoperatively
  Procedure performed in the Operating Room
Esophageal anastomotic leak not requiring surgery | Performed when clinically indicated up to 24 months postoperatively
  Barium swallow reports
Respiratory complications other than pneumonia | Performed when clinically indicated up to 24 months postoperatively
  Radiographic imaging reports

CONTACTS AND LOCATIONS:
Overall Officials: James Luketich, MD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - University of Pittsburgh Medical Center Presbyterian-Shadyside Hospital, Pittsburgh, Pennsylvania
  - Department of Cardiothoracic Surgery, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
Undecided

REFERENCES:
- [Derived] Luketich J, Sarkaria I, Levy R, Alicuben E, Gooding WE, Davis P, Awais O, Christie N, Levesque R, Ward J, Ryan J, Schuchert M, Pennathur A; University of Pittsburgh/UPMC MIE RAMIE Pyloroplasty Trial Study Group. A Phase III Randomized Controlled Trial of Pyloroplasty versus No Pyloroplasty in Patients Undergoing Minimally Invasive Esophagectomy or Robot-Assisted Minimally Invasive Esophagectomy. Ann Surg. 2025 Dec 19. doi: 10.1097/SLA.0000000000006997. Online ahead of print. PMID 41413794